CLINICAL TRIAL: NCT00809198
Title: The Effect of Kynex Versus Refresh Plus in Subjects With Mild to Moderate Dry Eye - A Parallel Group, Randomized, Masked Study
Brief Title: Kynex Versus Refresh Plus Study in Subject With Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RM-08-06
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Sodium Hyaluronate, Kynex, Carboxymethylcellulose sodium; Refresh Plus; Dry Eye; Cornea Staining; TBUT
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Hyaluronate (Experimental): Sodium Hyaluronate (Kynex)
  Interventions: Other: Sodium Hyaluronate
- Carboxymethylcellulose sodium (Active Comparator): Carboxymethylcellulose sodium (Refresh Plus)
  Interventions: Other: Carboxymethylcellulose sodium

INTERVENTIONS:
Other: Sodium Hyaluronate
  Other Names: Kynex
  Arms: Sodium Hyaluronate
Other: Carboxymethylcellulose sodium
  Other Names: Refresh Plus
  Arms: Carboxymethylcellulose sodium

SUMMARY:
The effect of Kynex versus Refresh Plus in subjects with mild to moderate dry eye.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older, of any race and either sex.
* Able to understand and sign an informed consent that has been approved by an Institutional Review Board.
* Criteria for the diagnosis must include the following two characteristics at Visit 1 (Day 1):
* Subjects' assessment of dry eye status (answer of at least "Some of the time" to the question, "How often have your eyes felt dry enough to want to use eye drops?"
* Sodium fluorescein (NaFl) corneal staining score sum of ≥3 in either eye (NEI scoring system).
* Able and willing to follow study instructions.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:
* History or evidence of ocular or intraocular surgery in either eye within the past three months.
* History of intolerance or hypersensitivity to any component of the study medications.
* History or evidence of epithelial herpes simplex keratitis (dendrictic keratitis); vaccine, active or recent varicella viral disease of the cornea and/or conjunctiva; ocular rosacea; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.
* Use of topical ocular medications during the study period.
* Subjects using systemic medications that may contribute to dry eye (e.g. cold and allergy medications, tricyclic antidepressants, hormone replacement therapies) may not be enrolled in the study unless they have been on a stable dosing regimen for a minimum of 30 days prior to Visit 1. In addition, the dosing regimen must remain stable throughout the study.
* Presence of ocular conditions such as active acute blepharitis, conjunctival infections, iritis, or any other ocular condition that may preclude the safe administration of the test article.
* Subjects unwilling to discontinue contact lens wear during the study period. Contact lens wear must have been discontinued at least one week prior to Visit 1.
* Current punctal occlusion of any type (e.g. collagen plugs, silicone plugs).
* Enrollment of the investigator or his or her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.
* Participation in any investigational drug or device study within 30 days of entering this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cornea Staining Score | 8 weeks

SECONDARY OUTCOMES:
Dry Eye and symptoms | 8 weeks